CLINICAL TRIAL: NCT03068910
Title: Study to Evaluate if Androgen-receptor Blockade (Spironolactone) Improves Progesterone-suppression of Wake Luteinizing Hormone Pulse Frequency in Pubertal Girls With Hyperandrogenism
Brief Title: Hyperandrogenemia and Altered Day-night LH Pulse Patterns
Acronym: CRM008
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Dr., MD, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18489; P50HD028934 (NIH)
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Hyperandrogenism; Polycystic Ovary Syndrome; Puberty
Keywords: Hyperandrogenism; Polycystic ovary syndrome; Puberty
MeSH Terms: conditions — Hyperandrogenism; Polycystic Ovary Syndrome | interventions — Progesterone; Spironolactone

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment allocation will be double-blinded. The blind will be broken in the event of substantial adverse effects that would also lead to study withdrawal. The blind for a given subject will be lifted after the subject completes the study and analysis is complete for that subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Experimental): Prior to the first or the second admission (randomly determined), participants will be pretreated for 2 weeks with spironolactone (50 mg twice daily).
  Interventions: Drug: Micronized progesterone; Drug: Placebo
- Placebo (Placebo Comparator): Prior to the first or the second admission (randomly determined), participants will be pretreated for 2 weeks with placebo (twice daily).
  Interventions: Drug: Spironolactone; Drug: Placebo

INTERVENTIONS:
Drug: Micronized progesterone — Micronized progesterone 0.8 mg/kg at 0700, 1500, 2300 and 0700 h. Progesterone is a natural hormone.
  Arms: Spironolactone
Drug: Spironolactone — Spironolactone is an androgen-receptor blocker commonly used (off-label) for hyperandrogenism. The spironolactone dose will be 50 mg taken orally twice daily (for two weeks before admission to the Clinical Research Unit).
  Arms: Placebo
Drug: Placebo — Placebo contains only inert ingredients and is not expected to exert any direct physiological effects.

SUMMARY:
The purpose of this study is to determine if, in mid- to late pubertal girls with hyperandrogenism, androgen-receptor blockade (spironolactone) improves the ability of progesterone to acutely reduce waking luteinizing hormone pulse frequency (primary endpoint).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded crossover study to test the following hypothesis: In mid- to late pubertal girls with hyperandrogenism (HA), acute progesterone suppression of waking LH pulse frequency is greater after 2 weeks of spironolactone pretreatment compared to after 2 weeks of placebo pretreatment. We will only study mid- to late pubertal girls with HA (i.e., girls who would be candidates for therapeutic spironolactone use). Subjects will complete two 18-hour Clinical Research Unit (CRU) admissions in separate menstrual cycles. Subjects will be randomized to be pretreated for 2 weeks with either oral spironolactone (50 mg twice daily) or placebo prior to the first CRU admission. Immediately before and during each CRU admission, oral micronized progesterone (0.8 mg/kg/dose) will be given at 0700, 1500, 2300, and 0700 h. During each CRU admission, blood will be obtained every 10 minutes through an indwelling iv catheter from 1800 to 1200 h. This will allow full characterization of pulsatile LH secretion in addition to other hormone measurements. Formal polysomnography will be performed during CRU admissions. A second CRU admission (performed at least 2 months later given blood withdrawal limits) will be identical to the first except that placebo pretreatment will exchanged for spironolactone pretreatment or vice versa (treatment crossover). The primary endpoint is LH pulse frequency while awake. (LH pulse frequency while asleep is an important secondary endpoint.) The wake LH pulse frequency data from the spironolactone and placebo admissions will be analyzed via a hierarchical linear mixed model (HLMM). The admission (spironolactone vs. placebo) will represent the fixed effect factor of the HLMM. Random effects will be utilized to account for the hierarchical variance-covariance structure of the two-period cross-over design. Wake LH pulse frequency in response to exogenous progesterone will be compared between the spironolactone admission and the placebo admission via a linear contrast of the HLMM least squares LH pulse frequency means. A similar analysis will be performed for sleep-related LH pulse frequency. Using published and preliminary data, we determined that, if 16 mid- to late pubertal girls with HA complete both admissions, we should have at least an 80% chance of detecting a 0.35 pulse/hour mean within-subject difference in wake LH pulse frequency between the spironolactone and placebo admissions with a two-sided false positive rejection rate of no more than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Mid- to late pubertal adolescent girl (at least Tanner breast stage 3, but no more than 2 years postmenarcheal)
* Hyperandrogenism, defined as a serum (calculated) free testosterone concentration greater than the Tanner stage-specific reference range and/or unequivocal evidence for hirsutism
* General good health (excepting overweight, obesity, hyperandrogenism, and adequately-treated hypothyroidism)
* Capable of and willing to provide informed assent (adolescents under age 16 years) and/or consent (adolescents over age 16 years; custodial parents or guardians of all adolescent volunteers)
* Willing to strictly avoid pregnancy with use of reliable non-hormonal methods during the study period

Exclusion Criteria:

* Inability/incapacity to provide informed consent
* Males will be excluded (hyperandrogenism is unique to females)
* Obesity resulting from a well-defined endocrinopathy or genetic syndrome
* Positive pregnancy test or current lactation
* Evidence for non-physiologic or non-PCOS causes of hyperandrogenism and/or anovulation
* Evidence of virilization (e.g., rapidly progressive hirsutism, deepening of the voice, clitoromegaly)
* Total testosterone > 150 ng/dl, which suggests the possibility of virilizing ovarian or adrenal tumor
* DHEA-S elevation > 1.5 times the upper reference range limit. Mild elevations may be seen in adolescent HA and in PCOS, and will be accepted in these groups.
* Early morning 17-hydroxyprogesterone > 200 ng/dl measured in the follicular phase, which suggests the possibility of congenital adrenal hyperplasia (if elevated during the luteal phase, the 17-hydroxyprogesterone will be repeated during the follicular phase). NOTE: If a 17-hydroxyprogesterone > 200 ng/dl is confirmed on repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl will be required for study participation.
* Abnormal thyroid stimulating hormone (TSH): Note that subjects with stable and adequately treated primary hypothyroidism, reflected by normal TSH values, will not be excluded.
* Hyperprolactinemia > 20% higher than the upper limit of normal. Mild prolactin elevations may be seen in adolescents and women with HA/PCOS, and elevations within 20% higher than the upper limit of normal will be accepted in this group.
* History and/or physical exam findings suggestive of Cushing's syndrome, adrenal insufficiency, or acromegaly
* History and/or physical exam findings suggestive of hypogonadotropic hypogonadism (e.g., symptoms of estrogen deficiency) including functional hypothalamic amenorrhea (which may be suggested by a constellation of symptoms including restrictive eating patterns, excessive exercise, psychological stress, etc.)
* Persistent hematocrit < 36% and hemoglobin < 12 g/dl.
* Severe thrombocytopenia (platelets < 50,000 cells/microliter) or leukopenia (total white blood count < 4,000 cells/microliter)
* Previous diagnosis of diabetes, fasting glucose > or = 126 mg/dl, or a hemoglobin A1c > or = 6.5%
* Persistent liver panel abnormalities, with two exceptions. Mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome. Also, mild transaminase elevations may be seen in obesity/HA/PCOS; therefore, elevations < 1.5 times the upper limit of normal will be accepted in this group.
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure, asthma requiring intermittent systemic corticosteroids, etc.)
* Decreased renal function evidenced by GFR < 60 ml/min/1.73m2
* A personal history of breast, ovarian, or endometrial cancer
* History of any other cancer diagnosis and/or treatment (with the exception of basal cell or squamous cell skin carcinoma) unless they have remained clinically disease free (based on appropriate surveillance) for five years
* History of allergy to micronized progesterone or spironolactone
* Body mass index (BMI)-for-age percentile < 5% (underweight)
* Due to the amount of blood being drawn, adolescent volunteers with body weight < 25 kg will be excluded.
* Restrictions on use of other drugs or treatments: No medications known to affect the reproductive system, glucose metabolism, lipid metabolism, or blood pressure can be taken in the 2 months prior to the screening visit and in the 3 months prior to the start of the study medications. Such medications include oral contraceptive pills, progestins, metformin, systemic glucocorticoids, some antipsychotic medications, and sympathomimetics/stimulants (e.g., methylphenidate).

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2016-07-21 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Luteinizing hormone (LH) pulse frequency | During first CRU admission and during the second CRU admission (which occurs at least 2 months after the first)
  LH pulse frequency while awake vs. while asleep

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, M.D., Principal Investigator — University of Virginia Center for Research in Reproduction
Locations (1):
- University of Virginia Clinical Research Unit, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share IPD. Data from this study will be deposited in the NICHD Data and Specimen Hub "DASH." We also plan to provide raw study data (de-identified) as supplementary materials in the resulting manuscript as was done for Kim SH, et al. Progesterone-mediated inhibition of the GnRH pulse generator: differential sensitivity as a function of sleep status. J Clin Endocrinol Metab 2018; 103: 1112-1121 [PMCID in process].